CLINICAL TRIAL: NCT00470197
Title: Phase I Study of a Pharmacologically Derived Hybrid Bolus-Infusion Schedule of Flavopiridol (NSC 649890, IND 46,211) Given in Timed Sequential Combination With Cytosine Arabinoside (Ara-C) and Mitoxantrone for Adults With Relapsed and Refractory Acute Leukemias
Brief Title: Flavopiridol, Cytarabine, and Mitoxantrone in Treating Patients With Relapsed or Refractory Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00243; NCI-2009-00243 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); J06133; CDR0000543443; J06133 (Other: Johns Hopkins University); 7889 (Other: CTEP); U01CA070095 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Malignant Neoplasm; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — alvocidib; Cytarabine; Mitoxantrone

ARMS (1):
- Arm I (Experimental): Patients receive flavopiridol IV over 30 minutes on days 1, 2, and 3. Patients receive cytarabine IV continuously over 72 hours beginning on day 6 and mitoxantrone hydrochloride IV over 60-120 minutes on day 9.
  Interventions: Drug: alvocidib; Drug: cytarabine; Drug: mitoxantrone hydrochloride; Other: pharmacological study

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone
Other: pharmacological study — Correlative study
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy, such as flavopiridol, cytarabine, and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving a new schedule of more than one drug (combination chemotherapy) may kill more cancer cells. This phase I trial is studying the side effects, best dose, and best schedule for flavopiridol when given together with cytarabine and mitoxantrone in treating patients with relapsed or refractory acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxicities of escalating doses of flavopiridol administered by "hybrid" bolus-infusion schedule and given in timed sequence with cytarabine and mitoxantrone hydrochloride in patients with refractory or relapsed acute leukemia.

II. Determine the incidence of clinical response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of flavopiridol. Patients receive flavopiridol IV over 30 minutes on days 1, 2, and 3.

Patients receive cytarabine IV continuously over 72 hours beginning on day 6 and mitoxantrone hydrochloride IV over 60-120 minutes on day 9. Treatment repeats every 35-63 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Serum and bone marrow samples are collected at baseline, during, and after completion of treatment for future studies. Flavopiridol levels are measured at baseline and on days 1-3 for pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed acute myeloid leukemia or acute lymphoblastic leukemia:

  * Relapsed >= 1 time OR refractory disease:

    * Patients who fail primary induction therapy or who relapse after achieving complete remission are eligible if they have received =< 3 prior courses of induction/reinduction therapy
* Relapsed >= 1 time OR refractory disease
* Patients who fail primary induction therapy or who relapse after achieving complete remission are eligible if they have received =< 3 prior courses of induction/reinduction therapy
* No active CNS leukemia
* ECOG performance status 0-2
* AST and ALT =< 5 times upper limit normal (ULN)
* Alkaline phosphatase =< 5 times ULN
* Bilirubin =< 2.0 mg/dL
* Creatinine =< 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* LVEF >= 45% by MUGA or ECHO
* No active, uncontrolled infection
* No other life-threatening illness
* No mental deficits and/or psychiatric history that would preclude study compliance
* No active graft-vs-host disease
* Recovered from all prior therapies
* At least 24 hours since prior hydroxyurea, steroids, imatinib mesylate, arsenic trioxide, interferon, or leukapheresis for blast count control
* At least 4 weeks since prior stem cell transplantation (autologous or allogeneic)
* At least 4 days since prior growth factors
* At least 3 weeks since prior chemotherapy, except for non-aplasia producing treatments (e.g., low-dose cyclophosphamide, hydroxyurea, interferon, imatinib mesylate, mercaptopurine, thalidomide, azacitidine, or decitabine)
* No prior flavopiridol
* No other concurrent chemotherapy, radiotherapy, or immunotherapy
* No acute promyelocytic leukemia (M3)
* No hyperleukocytosis with > 50,000 blasts/mm^3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-04; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by dose-limiting toxicities graded according to NCI-CTC version 3.0 | Up to 63 days

CONTACTS AND LOCATIONS:
Overall Officials: Judith Karp, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Karp JE, Smith BD, Resar LS, Greer JM, Blackford A, Zhao M, Moton-Nelson D, Alino K, Levis MJ, Gore SD, Joseph B, Carraway H, McDevitt MA, Bagain L, Mackey K, Briel J, Doyle LA, Wright JJ, Rudek MA. Phase 1 and pharmacokinetic study of bolus-infusion flavopiridol followed by cytosine arabinoside and mitoxantrone for acute leukemias. Blood. 2011 Mar 24;117(12):3302-10. doi: 10.1182/blood-2010-09-310862. Epub 2011 Jan 14. PMID 21239698